CLINICAL TRIAL: NCT05641792
Title: Continuous Glucose Monitoring for Emergency Laparotomy
Acronym: CLUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 420/2
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Peritonitis; Surgical Site Infection; Infections; Hyperglycemia; Hypoglycemia
Keywords: continuous glucose monitoring; CGM; Dexcom G6
MeSH Terms: conditions — Peritonitis; Surgical Wound Infection; Infections; Hyperglycemia; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM pre-, intra- and postoperatively (Experimental): Patients will have a Dexcom G6 system placed on admission on outer part of the arm, glycaemia will be monitored for 10 consecutive days
  Interventions: Device: CGM (Dexcom G6)

INTERVENTIONS:
Device: CGM (Dexcom G6) — Dexcom G6 system consists of a transmitter and sensor that measure interstitial glycaemia every 5 minutes. Measurements are transmitted via Bluetooth to a compatible device, that uploads the data on a virtual drive. This allows for remote real-time glycaemia monitoring on another device.
  Other Names: continuous glucose monitoring, CGM, Dexcom G6

SUMMARY:
CLUE trial aims to determine the feasibility and predictive value for surgical site infection (SSI) of continuous glucose monitoring (CGM) in emergency laparotomy patients with diffuse peritonitis.

DETAILED DESCRIPTION:
Hyperglycaemia commonly occurs during surgery due to a reaction to metabolic stress and trauma. It has been shown that improper glycemia control leads to impaired wound healing and a higher risk of other postoperative complications. Therefore, the investigators predict that number of hyperglycaemia episodes could be a predictor of SSI.

Continuous glucose monitoring allows for a minimally invasive real-time remote glycemia control, yet it has not been applied in an emergency surgery setting. Intraoperative glycemia monitoring would allow to determine the effect of specific interventions during a surgical procedure that may provoke hyperglycaemia.

CLUE is a single-centre prospective observational study held in an academic tertiary medical centre in Poland. Adult patients qualified for an emergency laparotomy for peritonitis in University Clinical Centre (UCC) Division of Oncological, Endocrine and General Surgery, with class ≥ III wounds according to Centers for Disease Control and Prevention (CDC) classification, will be eligible for the CLUE trial. Patients who will be unable or will refuse to express informed consent will be excluded. Patients will be co-enrolled in PRISTINE randomized health services study that aims to compare the effectiveness of negative pressure wound therapy (NPWT) and primary closure (PC) in surgical site infection prevention.

On admission day, patients will have a Dexcom G6 system placed on the outer part of the upper arm. Patients will undergo standard surgical procedures and perioperative care. Patients will be randomized to NPWT or PC according to PRISTINE protocol. Glycemia will be continuously monitored for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* emergency laparotomy for peritonitis
* written informed consent

Exclusion Criteria:

- open abdomen treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
feasibility of CGM system | 10 days
  measured as the drop-out rate caused by non-adherence of both patients and medical staff due to system detaching, problems with the receiving device (low battery. distance beyond Bluetooth communication range) etc.

SECONDARY OUTCOMES:
intra- and post-operative glycemia | 10 days
  number of hyperglycemia episodes
postoperative morbidity | 30 days
  all types of postoperative complications and their severity according to Clavien-Dindo scale (grade I to V; grade I represents any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention and grade 5 represents patient's death)
SSI rate | 30 days
  Surgical Site Infection according to Centre for Disease Control criteria:
  Infection occurring within the first 30 post-operative days with at least one of the following:
  * Purulent drainage from the incision
  * Organisms isolated from an aseptically obtained culture of fluid or tissue from the incision
  * Incision is deliberately opened by a surgeon AND at least one of the following signs/symptoms of infection:
    1. Pain or tenderness
    2. Localized swelling
    3. Redness
    4. Heat
  * Diagnosis of SSI by the surgeon or attending physician
  Due to the inability to implement CDC for wounds treated with NPWT, the investigators have included additional SSI criteria: the absolute necessity to prolong NPWT after 3rd day postop, an anergic wound morphology or slough.
effective wound closure | 30 days
  definitive wound closure, not followed by wound dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Spychalski, MD, PhD, Principal Investigator — MUG Division of General Surgery; Katarzyna Polomska, Principal Investigator — Medical University of Gdansk (MUG); Jaroslaw Kobiela, Prof., Principal Investigator — MUG Division of General Surgery
Locations (1):
- UCC Division of Oncological, Transplant and General Surgery, Gdansk, Pomeranian Voivodeship, Poland